CLINICAL TRIAL: NCT03121235
Title: PCR Based Detection of Azole Resistance in A. Fumigatus to Improve Patient Outcome. A Prospective Multicenter Observational Study.
Brief Title: PCR Based Detection of Azole Resistance in A. Fumigatus to Improve Patient Outcome.
Acronym: AzorMan
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Bart Rijnders, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2016-664
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Aspergillosis, Invasive Pulmonary
Keywords: aspergillosis; mycosis; neutropenia; hematologic diseases; AsperGenius PCR; Ambisome; Voriconazole
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Aspergillosis; Mycoses; Neutropenia; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Broncho-alveolar lavage specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: PCR based detection of azole resistance in A. fumigatus — Diagnosis and treatment of IA will be based on the results of a standardized diagnosis and treatment protocol that includes the use of the AsperGenius® PCR.

SUMMARY:
A standard treatment protocol for invasive aspergillosis (IA) will be implemented in several academic hematology centers in the Netherlands in which a diagnostic test demonstrating azole resistance by multiplex real-time polymerase chain reaction will guide the choice of appropriate antifungal treatment.

Objectives:

1. Improve the outcome of patients infected with azole resistant A. fumigatus by the early detection of Resistance Associated Mutations (RAMs) and with this the earlier initiation of the most appropriate therapy.
2. Monitor the prevalence of invasive aspergillosis due to strains carrying the TR34/L98H or the TR46/T289A/Y121F resistance associated mutations in the Netherlands.

DETAILED DESCRIPTION:
Invasive aspergillosis (IA) is the most common mould infection in immunocompromised haematological patients. A relatively low mortality is observed when diagnosis is made early and treatment with voriconazole, the first choice of treatment, is initiated promptly. However, azole resistance in Aspergillus fumigatus is increasingly reported in Europe. Fungal susceptibility testing is difficult, time consuming and not widely available. Furthermore, cultures remain negative in the majority of the patients with IA. AsperGenius®, is a CE certified multiplex real-time polymerase chain reaction (PCR) assay that allows for a simultaneous detection of the presence of Aspergillus species and identification of the most common mutations in the A. fumigatus CYP51A gene conferring resistance. The use of this PCR results in faster diagnosis of azole resistance and thus the initiation of appropriate therapy at an earlier point in time. A fast diagnosis and correct treatment leads to an improved outcome. After extensive discussions and a face-to-face meeting with 7 of the 8 UMC in the Netherlands a consensus diagnostic and therapeutic protocol was agreed upon. In this protocol, the AsperGenius® PCR will be used for the diagnosis of azole resistance and antifungal treatment will be changed if resistance is detected. This protocol is the current standard diagnostic and treatment approach at Erasmus MC.

Haematological patients suspected of having an invasive fungal pulmonary infection undergo BAL sampling as standard of care. AsperGenius® PCR on BAL sample allows to make a rapid diagnosis of invasive aspergillosis and gives information about azole resistance faster than standard time consuming methods like fungal culture and galactomannan measurement. A standard treatment protocol based on this new diagnostic tool is in place at Erasmus MC and will be implemented in the other study centres. The centres will be asked to send BAL sample of at least 1ml, preferably 2ml.

If RAMs are detected, the treating physician will be advised to switch from voriconazole to 1 of the following options:

1. Ambisome 3mg/kg IV
2. In case of treatment limiting toxicity of Ambisome IV, we suggest the use of an echinocandin in combination with posaconazole and aiming at serum Cthrough levels of 3-4mg/L
3. Step down therapy from IV therapy as described under 1 and 2 to oral therapy with posaconazole is allowed after at least 2 weeks of IV therapy and after a documented clinical and or radiological response. Posaconazole serum Cthrough levels of 3-4mg/L will be aimed for. Step down to posaconazole will not be done if an A. fumigatus strain with an MIC of >0.5 microgram/ml is cultured.
4. As an alternative to posaconazole step down, IV ambisome 5mg/kg thrice weekly can be given as well.

ELIGIBILITY:
Inclusion Criteria:

* Patient with underlying hematological disease
* Patient will undergo/underwent BAL sampling for suspected invasive fungal infection
* BAL samples should be submitted to the local microbiology lab for fungal culture and for galactomannan detection.
* The treating physician is planning to start voriconazole, isavuconazole or posaconazole after the BAL has been sampled while waiting for the culture or PCR results of the BAL sample or has already started voriconazole or posaconazole before BAL sampling.

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in this study:
* Antifungal therapy was started >120hours prior to BAL sampling (*)
* Antifungal prophylaxis with posaconazole or voriconazole for >5 days within the 2 weeks preceding BAL sampling
* Antifungal prophylaxis with itraconazole and at least half of the plasma itraconazole/hydroxy-itraconazole levels that were measured through therapeutic drug monitoring were above the minimum effective plasma concentration of 0.5mg/L (parental compound only, HLPC assay method). The minimum effective plasma concentration of 0.5mg/L for itraconazole has been established by the ECIL 6 meeting with a recommendation AII.

(*) Patients that develop new pulmonary infiltrates during antifungal prophylaxis (systemic azoles or aerosolized amphotericin B) can be included.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an underlying haematological disease (AML, CLL, CML, stem cell transplant etc.) aged 18 years and older are eligible if they are presenting with a new pulmonary infiltrate on chest CT-scan suspicious for invasive fungal infection and are planned to undergo or have undergone a bronchoscopic alveolar lavage (BAL).
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of antifungal treatment failure | 12 weeks
  Incidence of antifungal treatment failure in patients with the presence of RAM detected by the AsperGenius® resistance PCR. This incidence will be compared with a fixed failure rate set at 75%, based on the observed treatment failure in patients treated with voriconazole that were shown to carry azole resistant A. fumigatus.

SECONDARY OUTCOMES:
Demonstrate that early detection of azole resistance reduces the overall mortality. | 6 weeks
  This will be compared with a fixed mortality of 50%.
Demonstrate that a step down to oral posaconazole is a reasonable treatment option in patients that have responded to at least 2 weeks of IV antifungal therapy. | 12 weeks
  Posaconazole step down therapy will be considered effective if <35% of the patients treated with posaconazole oral monotherapy show progression of their invasive aspergillosis after documented response after at least 14 days of IV antifungal therapy.
Comparison of antifungal treatment failure in patients with the presence of RAM. | 24 weeks
  A group that received appropriate antifungal therapy soon will be compared with a group that received treatment late.

CONTACTS AND LOCATIONS:
Overall Officials: Bart JA Rijnders, MD/PhD, Principal Investigator — Internal Medicine and Infectious Diseases
Locations (8):
- Netherlands (8):
  - Academisch Medisch Centrum, Amsterdam
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht Universitair Medisch Centrum +, Maastricht
  - Radboud Medisch Universitair Centrum, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verweij PE, Zhang J, Debets AJM, Meis JF, van de Veerdonk FL, Schoustra SE, Zwaan BJ, Melchers WJG. In-host adaptation and acquired triazole resistance in Aspergillus fumigatus: a dilemma for clinical management. Lancet Infect Dis. 2016 Nov;16(11):e251-e260. doi: 10.1016/S1473-3099(16)30138-4. Epub 2016 Sep 13. PMID 27638360
- [Background] Vermeulen E, Maertens J, De Bel A, Nulens E, Boelens J, Surmont I, Mertens A, Boel A, Lagrou K. Nationwide Surveillance of Azole Resistance in Aspergillus Diseases. Antimicrob Agents Chemother. 2015 Aug;59(8):4569-76. doi: 10.1128/AAC.00233-15. Epub 2015 May 18. PMID 25987612
- [Background] van der Linden JW, Snelders E, Kampinga GA, Rijnders BJ, Mattsson E, Debets-Ossenkopp YJ, Kuijper EJ, Van Tiel FH, Melchers WJ, Verweij PE. Clinical implications of azole resistance in Aspergillus fumigatus, The Netherlands, 2007-2009. Emerg Infect Dis. 2011 Oct;17(10):1846-54. doi: 10.3201/eid1710.110226. PMID 22000354
- [Background] Chong GL, van de Sande WW, Dingemans GJ, Gaajetaan GR, Vonk AG, Hayette MP, van Tegelen DW, Simons GF, Rijnders BJ. Validation of a new Aspergillus real-time PCR assay for direct detection of Aspergillus and azole resistance of Aspergillus fumigatus on bronchoalveolar lavage fluid. J Clin Microbiol. 2015 Mar;53(3):868-74. doi: 10.1128/JCM.03216-14. Epub 2015 Jan 7. PMID 25568431
- [Background] Verweij PE, Chowdhary A, Melchers WJ, Meis JF. Azole Resistance in Aspergillus fumigatus: Can We Retain the Clinical Use of Mold-Active Antifungal Azoles? Clin Infect Dis. 2016 Feb 1;62(3):362-8. doi: 10.1093/cid/civ885. Epub 2015 Oct 20. PMID 26486705
- [Background] Mavridou E, Bruggemann RJ, Melchers WJ, Mouton JW, Verweij PE. Efficacy of posaconazole against three clinical Aspergillus fumigatus isolates with mutations in the cyp51A gene. Antimicrob Agents Chemother. 2010 Feb;54(2):860-5. doi: 10.1128/AAC.00931-09. Epub 2009 Nov 16. PMID 19917751
- [Background] Verweij PE, Ananda-Rajah M, Andes D, Arendrup MC, Bruggemann RJ, Chowdhary A, Cornely OA, Denning DW, Groll AH, Izumikawa K, Kullberg BJ, Lagrou K, Maertens J, Meis JF, Newton P, Page I, Seyedmousavi S, Sheppard DC, Viscoli C, Warris A, Donnelly JP. International expert opinion on the management of infection caused by azole-resistant Aspergillus fumigatus. Drug Resist Updat. 2015 Jul-Aug;21-22:30-40. doi: 10.1016/j.drup.2015.08.001. Epub 2015 Aug 7. PMID 26282594
- [Background] Verweij PE, Lestrade PP, Melchers WJ, Meis JF. Azole resistance surveillance in Aspergillus fumigatus: beneficial or biased? J Antimicrob Chemother. 2016 Aug;71(8):2079-82. doi: 10.1093/jac/dkw259. PMID 27494831
- [Background] Chong GM, van der Beek MT, von dem Borne PA, Boelens J, Steel E, Kampinga GA, Span LF, Lagrou K, Maertens JA, Dingemans GJ, Gaajetaan GR, van Tegelen DW, Cornelissen JJ, Vonk AG, Rijnders BJ. PCR-based detection of Aspergillus fumigatus Cyp51A mutations on bronchoalveolar lavage: a multicentre validation of the AsperGenius assay(R) in 201 patients with haematological disease suspected for invasive aspergillosis. J Antimicrob Chemother. 2016 Dec;71(12):3528-3535. doi: 10.1093/jac/dkw323. Epub 2016 Aug 15. PMID 27530755